CLINICAL TRIAL: NCT01728584
Title: Randomized, Controlled, Parallel-Group, Double-Blind Trial to Compare the Use of Deep or Standard Neuromuscular Blockade in Combination With Low or Standard Insufflation Pressures Using a 2x2 Factorial Design in Patients Undergoing Laparoscopic Cholecystectomy (Protocol No. MK-8616-076-03 Also Known as SCH 900616, P07982)
Brief Title: A Study Comparing the Use of Deep or Standard Neuromuscular Blockade in Combination With Low or Standard Insufflation Pressures in Participants Undergoing Laparoscopic Cholecystectomy (P07982)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P07982; MK-8616-076 (Other: Merck); 2012-001886-33 (EudraCT Number)
Record Dates: First submitted 2012-10-16; First posted 2012-11-20 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Gallbladder Disease
MeSH Terms: conditions — Gallbladder Diseases | interventions — Rocuronium; Insufflation; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard NMB and Standard Insufflation Pressure (Experimental): Treatment condition for this arm is Standard NMB (depth of blockade at a targeted Train of Four [TOF] ratio of 10%)/Standard insufflation pressure (starting pressure of 12 mmHg).
  Interventions: Drug: Rocuronium; Other: Insufflation; Drug: Sugammadex
- Standard NMB and Low Insufflation Pressure (Experimental): Treatment condition for this arm is Standard NMB (depth of blockade at a targeted TOF ratio of 10%)/Low insufflation pressure (starting pressure of 8 mmHg).
  Interventions: Drug: Rocuronium; Other: Insufflation; Drug: Sugammadex
- Deep NMB and Standard Insufflation Pressure (Experimental): Treatment condition for this arm is Deep NMB (depth of blockade of 1-2 PTCs)/Standard insufflation pressure (starting pressure of 12 mmHg).
  Interventions: Drug: Rocuronium; Other: Insufflation; Drug: Sugammadex
- Deep NMB and Low Insufflation Pressure (Experimental): Treatment condition for this arm is Deep NMB (depth of blockade of 1-2 PTCs)/Low insufflation pressure (starting pressure of 8 mmHg).
  Interventions: Drug: Rocuronium; Other: Insufflation; Drug: Sugammadex

INTERVENTIONS:
Drug: Rocuronium — NMB will be induced by intravenous (IV) administration of a bolus dose of 0.45 mg/kg rocuronium. NMB will be maintained using rocuronium infusion or additional bolus doses as needed for the management of NMB to the targeted depth according to the assigned treatment condition. - Standard NMB - administration of neuromuscular blocking agent (NMBA) titrated to a depth of blockade at a targeted TOF ratio of 10% (range: TOF count 2-3 to TOF ratio of 20%). - Deep NMB - administration of NMBA titrated to a targeted depth of 1-2 Post Tetanic Counts (PTCs) (range: 1-5 PTC).
  Other Names: Zemuron® Injection (rocuronium bromide)
Other: Insufflation — Insufflation (injection) of carbon dioxide will be used to induce pneumoperitoneum, which is presence of air or gas in the abdominal (peritoneal) cavity.
  * Standard insufflation pressure - a starting pressure of 12 mmHg will be used.
  * Low insufflation pressure - a starting pressure of 8 mmHg will be used.
Drug: Sugammadex — NMB will be reversed with IV administration of 2 or 4 mg/kg sugammadex (depending on the depth of NMB) according to the approved label for sugammadex.
  Other Names: sugammadex sodium injection; SCH 900616; Org 25969; Bridion®

SUMMARY:
The purpose of this pilot study is to compare the use of deep or standard neuromuscular blockade (NMB) in combination with low or standard insufflation pressure in participants undergoing a surgical procedure, laparoscopic cholecystectomy. Insufflation refers to the injection of carbon dioxide into the abdomen during the laparoscopic surgery, to allow visualization of and access to the surgical field. The primary hypothesis of the study is that the use of sustained deep NMB improves the surgeon's overall satisfaction with surgical conditions as compared to standard NMB. The in-patient surgery is performed on Day 1 and the participant remains hospitalized for at least 48 hours following the surgery (or at least 24 hours following the surgery, if local practice does not allow 48 hours of hospitalization post surgery). On Day 8, a follow-up visit/contact including all participants occurs.

DETAILED DESCRIPTION:
During procedure, surgeon (who was blinded to random assignment) could request that unblinded anesthetist change the randomized treatment conditions (called a "rescue intervention"), if surgeon considered surgical conditions to be unacceptable. This was to be done systematically as follows: If the participant is on standard NMB, the preferred rescue intervention should be to increase the NMB to a depth of 1-2 PTCs; for such a participant the second option (if participant is also on low insufflation pressure) should be the increase of insufflation pressure by 4 mmHg. If the participant is already on deep NMB, the preferred option should be (if participant is also on low insufflation pressure) the increase of insufflation pressure by 4 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class 1 or 2 or 3
* Scheduled to undergo an elective in-patient laparoscopic cholecystectomy procedure under general anesthesia with total intravenous anesthesia (TIVA) using propofol and remifentanil
* Eligible to undergo rocuronium-induced NMB for endotracheal intubation and maintenance of NMB
* Will recover in the post-anesthesia care unit (PACU) and remain in the hospital for at least 48 hours following the surgical procedure (or at least 24 hours following the surgical procedure, if local practice does not allow 48 hours of hospitalization post surgery)
* Body mass index (BMI) ≤35
* Willing and able to adhere to visit schedules including all required study assessments on Day 3 through 8 (daily pain and medication diary entry)
* For sexually active female participants of child-bearing potential - able to use a medically accepted method of contraception through 7 days after receiving protocol-specified medication

Exclusion criteria:

* Neuromuscular disorders that may affect NMB and/or trial assessments
* Lifetime history of previous abdominal surgery, including laparotomies, Cesarean section, laparoscopic procedures or diagnostic laparoscopies
* Substance abuse or dependence (excluding nicotine) within the past 6 months
* History of a chronic pain condition (requiring continuous/daily pain medication prior to surgery)
* For female participants - lifetime history of a Cesarean section, or has given birth to one or more children within the last year, or is currently pregnant or has the intention to become pregnant between randomization and pregnancy follow-up contact ≥30 days after administration of trial treatments (rocuronium, sugammadex)
* Evidence of acute cholecystitis
* Dialysis-dependency or suspected of having severe renal insufficiency
* Significant hepatic dysfunction that would prevent participation in the trial
* History of or family history of malignant hyperthermia
* Allergy to trial treatments (rocuronium or sugammadex) or their excipients, to opioids/opiates, or other medication used during general anesthesia
* Received or is planned to receive toremifene or fusidic acid within 24 hours before or after receiving rocuronium or sugammadex
* Expected transfer to an Intensive Care Unit after surgery
* Any clinically significant condition or situation, other than the reason for the cholecystectomy that would interfere with the trial evaluations or optimal participation in the trial
* Used any investigational drugs within 30 days of randomization
* Participated in any other clinical trial within 30 days of signing the informed consent form of the current trial
* Participated in any other clinical trial involving any personnel of the investigational or Sponsor staff directly involved with this trial
* Is a family member of any personnel of the investigational or Sponsor staff directly involved with this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2014-04-29 (Actual); Study Completion 2014-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- Merck Sharp & Dohme GmbH, Haar, Germany
- MSD Italia S.r.l., Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rosenberg J, Herring WJ, Blobner M, Mulier JP, Rahe-Meyer N, Woo T, Li MK, Grobara P, Assaid CA, Fennema H, Szegedi A. Deep Neuromuscular Blockade Improves Laparoscopic Surgical Conditions: A Randomized, Controlled Study. Adv Ther. 2017 Apr;34(4):925-936. doi: 10.1007/s12325-017-0495-x. Epub 2017 Mar 1. PMID 28251555

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 4 arms based on combinations of neuromuscular blockade (NMB) depth and insufflation pressure level. During procedure, blinded surgeon could request that unblinded anesthetist change the randomized treatment conditions ("rescue intervention"), if surgeon considered surgical conditions to be unacceptable.
Groups:
- Standard NMB and Standard Insufflation Pressure: Treatment condition for this reporting group is Standard (Std) NMB (depth of blockade at a targeted Train of Four [TOF] ratio of 10%)/Standard insufflation pressure (starting pressure of 12 mmHg).
- Standard NMB and Low Insufflation Pressure: Treatment condition for this reporting group is Standard NMB (depth of blockade at a targeted TOF ratio of 10%)/Low insufflation pressure (starting pressure of 8 mmHg).
- Deep NMB and Standard Insufflation Pressure: Treatment condition for this reporting group is Deep NMB (depth of blockade of 1-2 Post Tetanic Counts [PTCs])/Standard insufflation pressure (starting pressure of 12 mmHg).
- Deep NMB and Low Insufflation Pressure: Treatment condition for this reporting group is Deep NMB (depth of blockade of 1-2 PTCs)/Low insufflation pressure (starting pressure of 8 mmHg).
Period: Overall Study
Arm/Group | Standard NMB and Standard Insufflation Pressure | Standard NMB and Low Insufflation Pressure | Deep NMB and Standard Insufflation Pressure | Deep NMB and Low Insufflation Pressure
Started | 36 (Randomized) | 30 (Randomized - NMB/pressure conditions were changed in 7 (2 to Std/Std, 4 to Deep/Std, 1 to Deep/Low)) | 31 (Randomized) | 30 (Randomized - NMB/pressure conditions were changed in 5 (all to Deep/Std))
Completed | 28 | 30 | 30 | 29
Not Completed | 8 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Screen failure | 1 | 0 | 0 | 0
Not completed — Other reason (not specified) | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants as randomized
Groups:
- Standard NMB and Standard Insufflation Pressure: Treatment condition for this reporting group is Standard NMB (depth of blockade at a targeted TOF ratio of 10%)/Standard insufflation pressure (starting pressure of 12 mmHg).
- Deep NMB and Standard Insufflation Pressure: Treatment condition for this reporting group is Deep NMB (depth of blockade of 1-2 PTCs)/Standard insufflation pressure (starting pressure of 12 mmHg).
- Total: Total of all reporting groups
Arm/Group | Standard NMB and Standard Insufflation Pressure | Standard NMB and Low Insufflation Pressure | Deep NMB and Standard Insufflation Pressure | Deep NMB and Low Insufflation Pressure | Total
Number analyzed (Participants) | 36 | 30 | 31 | 30 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (17.7) | 39.1 (13.6) | 43.5 (15.6) | 46.7 (13.8) | 43.9 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 13 | 9 | 48
  Male | 21 | 19 | 18 | 21 | 79

OUTCOME MEASURES:

1. Primary Outcome: Score on Surgeon's Assessment of Overall Satisfaction With the Surgical Conditions: By Depth of NMB (Standard, Deep) and Insufflation Pressure (Standard, Low)
Description: At the end of the procedure the surgeon responds to the following question, using an 11-point scale from 0 (poor, needed intervention) to 10 (excellent): "How satisfied were you overall with the surgical conditions related to anesthesia and pneumoperitoneum during the surgery you just performed?" If at any time the surgeon requests a rescue intervention, the overall assessment of surgical conditions should be rated as 0 (=poor, needed intervention). The surgeon will rate the surgical conditions according to his opinion but if a rescue intervention has been applied, that individual participant will be counted with a score of zero in the analysis.
Time Frame: End of surgery (Day 1)
Population: Randomized participants with available data who had NMB and pneumoperitoneum for laparoscopic surgery, and did not convert to open surgery before NMB and/or pressure application. Participants were included in the treatment arm to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Standard NMB: Treatment condition for this reporting group is Standard NMB (depth of blockade at a targeted TOF ratio of 10%), whether in combination with Standard or Low insufflation pressure. Therefore, the included arms are Standard NMB/Standard insufflation pressure and Standard NMB/Low insufflation pressure.
- Deep NMB: Treatment condition for this reporting group is Deep NMB (depth of blockade of 1-2 PTCs), whether in combination with Standard or Low insufflation pressure. Therefore, the included arms are Deep NMB/Standard insufflation pressure and Deep NMB/Low insufflation pressure.
- Standard Insufflation Pressure: Treatment condition for this reporting group is Standard insufflation pressure (starting pressure of 12 mmHg), whether in combination with Standard or Deep NMB. Therefore, the included arms are Standard NMB/Standard insufflation pressure and Deep NMB/Standard insufflation pressure.
- Low Insufflation Pressure: Treatment condition for this reporting group is Low insufflation pressure (starting pressure of 8 mmHg), whether in combination with Standard or Deep NMB. Therefore, the included arms are Standard NMB/Low insufflation pressure and Deep NMB/Low insufflation pressure.
Arm/Group | Standard NMB | Deep NMB | Standard Insufflation Pressure | Low Insufflation Pressure
Number analyzed (Participants) | 60 | 60 | 60 | 60
score on a scale | 6.83 [5.97 to 7.69] | 7.92 [7.05 to 8.80] | 8.89 [8.05 to 9.72] | 5.87 [4.96 to 6.77]
Statistical Analysis 1: Comparison: Standard NMB vs Deep NMB; Primary hypothesis - deep NMB improves surgeon's overall satisfaction with the surgical conditions compared to standard NMB; Test type: Superiority or Other; p = 0.026, ANCOVA; Analysis of covariance (ANCOVA) model included factors depth of NMB, level of pressure, surgeon and body mass index (BMI); Difference in Least Squares (LS) Means = 1.09, 95% CI 2-sided [0.13 to 2.04] — Difference is deep versus standard NMB
Statistical Analysis 2: Comparison: Standard Insufflation Pressure vs Low Insufflation Pressure; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Difference in LS Means = -3.02, 95% CI 2-sided [-3.99 to -2.05] — Difference is low versus standard pressure

2. Primary Outcome: Score on Surgeon's Assessment of Overall Satisfaction With the Surgical Conditions: By Treatment Arm
Description: as for outcome 1
Time Frame: End of surgery (Day 1)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a acale
Arm/Group | Standard NMB and Standard Insufflation Pressure | Standard NMB and Low Insufflation Pressure | Deep NMB and Standard Insufflation Pressure | Deep NMB and Low Insufflation Pressure
Number analyzed (Participants) | 30 | 30 | 30 | 30
score on a acale | 8.65 [7.58 to 9.72] | 4.99 [3.88 to 6.11] | 9.09 [8.82 to 10.17] | 6.69 [5.57 to 7.80]
Statistical Analysis 1: Comparison: Standard NMB and Standard Insufflation Pressure vs Standard NMB and Low Insufflation Pressure; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Test type: Superiority or Other; Difference in Least Squares (LS) Means = 3.66, 95% CI 2-sided [2.30 to 5.02] — Difference is standard NMB/standard pressure versus standard NMB/low pressure
Statistical Analysis 2: Comparison: Standard NMB and Standard Insufflation Pressure vs Deep NMB and Standard Insufflation Pressure; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Test type: Superiority or Other; Difference in LS Means = -0.44, 95% CI 2-sided [-1.80 to 0.91] — Difference is standard NMB/standard pressure versus deep NMB/standard pressure
Statistical Analysis 3: Comparison: Standard NMB and Standard Insufflation Pressure vs Deep NMB and Low Insufflation Pressure; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Test type: Superiority or Other; Difference in LS Means = 1.96, 95% CI 2-sided [0.57 to 3.36] — Difference is standard NMB/standard pressure versus deep NMB/low pressure
Statistical Analysis 4: Comparison: Standard NMB and Low Insufflation Pressure vs Deep NMB and Standard Insufflation Pressure; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Test type: Superiority or Other; Difference in LS Means = -4.10, 95% CI 2-sided [-5.42 to -2.78] — Difference is standard NMB/low pressure versus deep NMB/standard pressure
Statistical Analysis 5: Comparison: Standard NMB and Low Insufflation Pressure vs Deep NMB and Low Insufflation Pressure; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Test type: Superiority or Other; Difference in LS Means = -1.70, 95% CI 2-sided [-3.01 to -0.38] — Difference is standard NMB/low pressure versus deep NMB/low pressure
Statistical Analysis 6: Comparison: Deep NMB and Standard Insufflation Pressure vs Deep NMB and Low Insufflation Pressure; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Test type: Superiority or Other; Difference in LS Means = 2.41, 95% CI 2-sided [1.08 to 3.74] — Difference is deep NMB/standard pressure versus deep NMB/low pressure

3. Secondary Outcome: Participant's Overall Average Pain Score in the First 24 Hours After Administration of Sugammadex: By Depth of NMB (Standard, Deep) and Insufflation Pressure (Standard, Low)
Description: Participants rated pain at 1, 2, 4, 24 and 48 hours after the administration of sugammadex on day of surgery (Day 1), and daily from Day 3 to Day 8. Pain rating was made using an 11-point scale from 0 (no pain) to 10 (severe pain). Separate ratings were made for overall pain at rest, pain when provoked (e.g., due to participant transition from lying to sitting position) and shoulder pain at rest. The participant's overall average pain score within 24 hours after sugammadex was the average of all pain assessments (including all 3 pain types assessed) at 1, 2, 4 and 24 hours after sugammadex dose.
Time Frame: Up to 24 hours after administration of sugammadex on Day 1
Population: Randomized participants with available data who had NMB or pneumoperitoneum for laparoscopic surgery, or received sugammadex, and did not convert to open surgery before NMB and/or pressure. Participants were included in arm corresponding to treatment actually received, which in case of rescue intervention was the post-intervention condition.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard NMB | Deep NMB | Standard Insufflation Pressure | Low Insufflation Pressure
Number analyzed (Participants) | 55 | 65 | 71 | 49
score on a scale | 2.48 [2.02 to 2.93] | 2.83 [2.39 to 3.28] | 2.74 [2.34 to 3.15] | 2.57 [2.07 to 3.07]
Statistical Analysis 1: Comparison: Standard NMB vs Deep NMB; Test type: Superiority or Other; p = 0.148, ANOVA; Analysis of variance (ANOVA) model included factors depth of NMB, level of pressure, gender and surgeon; Difference in LS Means = 0.35, 95% CI 2-sided [-0.13 to 0.84] — Difference is deep versus standard NMB
Statistical Analysis 2: Comparison: Standard Insufflation Pressure vs Low Insufflation Pressure; Key secondary hypothesis - low insufflation pressure improves overall average pain score in first 24 hours compared to standard insufflation pressure; Test type: Superiority or Other; p = 0.494, ANOVA — To control for multiple testing, this difference was formally tested only if comparison of surgeon's overall satisfaction with surgical conditions for deep versus standard NMB was significant at the 5% level, with greater satisfaction for deep NMB; ANOVA model included factors depth of NMB, level of pressure, gender and surgeon; Difference in LS Means = -0.17, 95% CI 2-sided [-0.67 to 0.33] — Difference is low versus standard pressure

4. Secondary Outcome: Participant's Overall Average Pain Score in the First 24 Hours After Administration of Sugammadex: By Treatment Arm
Description: as for outcome 3
Time Frame: Up to 24 hours after administration of sugammadex on Day 1
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard NMB and Standard Insufflation Pressure | Standard NMB and Low Insufflation Pressure | Deep NMB and Standard Insufflation Pressure | Deep NMB and Low Insufflation Pressure
Number analyzed (Participants) | 32 | 23 | 39 | 26
score on a scale | 2.42 [1.90 to 2.93] | 2.62 [1.98 to 3.26] | 3.06 [2.56 to 3.57] | 2.57 [1.97 to 3.17]
Statistical Analysis 1: Comparison: Standard NMB and Standard Insufflation Pressure vs Standard NMB and Low Insufflation Pressure; ANOVA model included factors treatment group, gender and surgeon; Test type: Superiority or Other; Difference in LS Means = -0.20, 95% CI 2-sided [-0.92 to 0.52] — Difference is standard NMB/standard pressure versus standard NMB/low pressure
Statistical Analysis 2: Comparison: Standard NMB and Standard Insufflation Pressure vs Deep NMB and Standard Insufflation Pressure; ANOVA model included factors treatment group, gender and surgeon; Test type: Superiority or Other; Difference in LS Means = -0.65, 95% CI 2-sided [-1.27 to -0.02] — Difference is standard NMB/standard pressure versus deep NMB/standard pressure
Statistical Analysis 3: Comparison: Standard NMB and Standard Insufflation Pressure vs Deep NMB and Low Insufflation Pressure; ANOVA model included factors treatment group, gender and surgeon; Test type: Superiority or Other; Difference in LS Means = -0.15, 95% CI 2-sided [-0.84 to 0.53] — Difference is standard NMB/standard pressure versus deep NMB/low pressure
Statistical Analysis 4: Comparison: Standard NMB and Low Insufflation Pressure vs Deep NMB and Standard Insufflation Pressure; ANOVA model included factors treatment group, gender and surgeon; Test type: Superiority or Other; Difference in LS Means = -0.45, 95% CI 2-sided [-1.15 to 0.26] — Difference is standard NMB/low pressure versus deep NMB/standard pressure
Statistical Analysis 5: Comparison: Standard NMB and Low Insufflation Pressure vs Deep NMB and Low Insufflation Pressure; ANOVA model included factors treatment group, gender and surgeon; Test type: Superiority or Other; Difference in LS Means = 0.05, 95% CI 2-sided [-0.69 to 0.78] — Difference is standard NMB/low pressure versus deep NMB/low pressure
Statistical Analysis 6: Comparison: Deep NMB and Standard Insufflation Pressure vs Deep NMB and Low Insufflation Pressure; ANOVA model included factors treatment group, gender and surgeon; Test type: Superiority or Other; Difference in LS Means = 0.49, 95% CI 2-sided [-0.17 to 1.16] — Difference is deep NMB/standard pressure versus deep NMB/low pressure

5. Secondary Outcome: Score on Surgeon's Assessment of Overall Satisfaction With the Visibility of the Surgical Field: By Depth of NMB (Standard, Deep)
Description: At the end of the procedure the surgeon responds to the following question, using an 11-point scale from 0 (poor, unacceptable visibility) to 10 (excellent): "How satisfied were you overall with the visual field during the surgery you just performed?" If at any time the surgeon requests a rescue intervention, the surgeon will rate his overall satisfaction with the visibility of the surgical field according to his opinion, but if a rescue intervention has been applied, that individual participant will be counted with a score of zero in the analysis.
Time Frame: End of surgery (Day 1)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard NMB | Deep NMB
Number analyzed (Participants) | 60 | 60
score on a scale | 6.88 [6.02 to 7.75] | 7.80 [6.92 to 8.68]
Statistical Analysis 1: Comparison: Standard NMB vs Deep NMB; Test type: Superiority or Other; p = 0.063, ANCOVA — Not controlled for multiple testing; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Difference in LS Means = 0.91, 95% CI 2-sided [-0.05 to 1.87] — Difference is deep versus standard NMB

6. Secondary Outcome: Score on Surgeon's Assessment of the Overall Adequacy of Muscle Relaxation During Surgery: By Depth of NMB (Standard, Deep)
Description: At the end of the procedure the surgeon responds to the following question, using an 11-point scale from 0 (poor, unacceptable muscle relaxation, required intervention) to 10 (excellent): "How do you rate the overall adequacy of muscle relaxation during the surgery you just performed?"
Time Frame: End of surgery (Day 1)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard NMB | Deep NMB
Number analyzed (Participants) | 60 | 60
score on a scale | 8.05 [7.56 to 8.54] | 8.87 [8.37 to 9.37]
Statistical Analysis 1: Comparison: Standard NMB vs Deep NMB; Test type: Superiority or Other; p = 0.004, ANCOVA — Not controlled for multiple testing; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Difference in LS Means = 0.82, 95% CI 2-sided [0.27 to 1.37] — Difference is deep versus standard NMB

7. Secondary Outcome: Score on Surgeon's Assessment of the Overall Adequacy of Insufflation Pressure During Surgery: By Depth of NMB (Standard, Deep)
Description: At the end of the procedure the surgeon responds to the following question, using an 11-point scale from 0 (poor, unacceptable insufflation pressure, required intervention) to 10 (excellent): "How do you rate the overall adequacy of insufflation pressure during the surgery you just performed?"
Time Frame: End of surgery (Day 1)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard NMB | Deep NMB
Number analyzed (Participants) | 60 | 60
score on a scale | 6.73 [6.01 to 7.45] | 7.86 [7.12 to 8.59]
Statistical Analysis 1: Comparison: Standard NMB vs Deep NMB; Test type: Superiority or Other; p = 0.006, ANCOVA — Not controlled for multiple testing; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Difference in LS Means = 1.12, 95% CI 2-sided [0.32 to 1.92] — Difference is deep versus standard NMB

8. Secondary Outcome: Number of Times Participant's Movements or Increased Muscle Tone Interfered With the Surgical Conditions During Laparoscopy: By Depth of NMB (Standard, Deep)
Description: At the end of the procedure the surgeon responds to the following question: "How many times did patient's movements (coughing, bucking, hiccup) or increased muscle tone (resistance, difficulty to close fasciae or skin) interfere with your surgery?"
Time Frame: During surgery, approximate duration of 1-2 hours (Day 1)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: instances of occurrence that interfered
Arm/Group | Standard NMB | Deep NMB
Number analyzed (Participants) | 60 | 59
instances of occurrence that interfered | 0.92 [0.33 to 1.52] | 0.32 [-0.29 to 0.92]
Statistical Analysis 1: Comparison: Standard NMB vs Deep NMB; Test type: Superiority or Other; p = 0.073, ANCOVA — Not controlled for multiple testing; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Difference in LS Means = -0.61, 95% CI 2-sided [-1.27 to 0.06] — Difference is deep versus standard NMB

9. Secondary Outcome: Score on Surgeon's Assessment of the Effect Participant's Movements During Surgery Had on the Overall Surgical Procedure: By Depth of NMB (Standard, Deep)
Description: At the end of the procedure the surgeon responds to the following question, using an 11-point scale from 0 (extremely disruptive) to 10 (not disruptive): "How did the patient movements described above disrupt your surgical performance?" This refers to participant movements during surgery.
Time Frame: End of surgery (Day 1)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard NMB | Deep NMB
Number analyzed (Participants) | 60 | 60
score on a scale | 9.21 [8.72 to 9.70] | 9.94 [9.45 to 10.44]
Statistical Analysis 1: Comparison: Standard NMB vs Deep NMB; Test type: Superiority or Other; p = 0.009, ANCOVA — Not controlled for multiple testing; ANCOVA model included factors depth of NMB, level of pressure, surgeon and BMI; Difference in LS Means = 0.74, 95% CI 2-sided [0.19 to 1.28] — Difference is deep versus standard NMB

10. Secondary Outcome: Number of Participants With Rescue Actions Performed During Surgery in Order to Improve Insufficient Surgical Conditions: By Treatment Arm
Description: During procedure, surgeon (who was blinded to random assignment) could request that unblinded anesthetist change the randomized treatment conditions (called a "rescue intervention"), if surgeon considered surgical conditions to be unacceptable. This was to be done systematically as follows: If the participant is on standard NMB, the preferred rescue intervention should be to increase the NMB to a depth of 1-2 PTCs; for such a participant the second option (if participant is also on low insufflation pressure) should be the increase of insufflation pressure by 4 mm Hg. If the participant is already on deep NMB, the preferred option should be (if participant is also on low insufflation pressure) the increase of insufflation pressure by 4 mm Hg. The unblinded anesthetist recorded any rescue actions performed. This measure presents the number of participants: with any rescue action performed, with rescue change in depth of NMB, with rescue change in insufflation pressure level.
Time Frame: During surgery, approximate duration of 1-2 hours (Day 1)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Standard NMB and Standard Insufflation Pressure | Standard NMB and Low Insufflation Pressure | Deep NMB and Standard Insufflation Pressure | Deep NMB and Low Insufflation Pressure
Number analyzed (Participants) | 31 | 30 | 31 | 30
participants
  Number with rescue action performed | 0 | 7 | 0 | 5
  Number with rescue change in depth of NMB | 0 | 5 | 0 | 0
  Number with rescue change in pressure level | 0 | 6 | 0 | 5

11. Secondary Outcome: Participant's Daily Assessment of Overall Pain at Rest During Post Operative Period: By Treatment Arm
Description: Participants rated pain at 1, 2, 4, 24 and 48 hours after the administration of sugammadex on day of surgery (Day 1), and daily (in the morning) from Day 3 to Day 8. Pain rating was made using an 11-point scale from 0 (no pain) to 10 (severe pain). Separate ratings were made for overall pain at rest, pain when provoked (e.g., due to participant transition from lying to sitting position) and shoulder pain at rest. This measure summarizes the assessment of overall pain at rest for the study days following the surgery.
Time Frame: Days 2 to 8
Population: Randomized participants with available data who had NMB or pneumoperitoneum for laparoscopic surgery, or received sugammadex. Participants were included in arm corresponding to treatment actually received, which in case of rescue intervention was the post-intervention condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard NMB and Standard Insufflation Pressure | Standard NMB and Low Insufflation Pressure | Deep NMB and Standard Insufflation Pressure | Deep NMB and Low Insufflation Pressure
Number analyzed (Participants) | 33 | 23 | 40 | 26
score on a scale
  24 hours after sugammadex dose (n=29, 22, 38, 25) | 1.66 (1.45) | 2.23 (2.09) | 2.24 (1.62) | 2.48 (2.20)
  48 hours after sugammadex dose (n=27, 22, 33, 23) | 1.22 (1.45) | 1.41 (1.68) | 1.73 (1.53) | 1.83 (1.64)
  Day 3 (N=22, 20, 30, 17) | 0.86 (0.89) | 1.65 (1.76) | 1.87 (1.59) | 2.00 (1.84)
  Day 4 (N=28, 20, 37, 23) | 0.89 (1.23) | 1.05 (1.50) | 1.76 (1.55) | 1.04 (1.46)
  Day 5 (N=27, 21, 38, 24) | 0.89 (1.01) | 1.00 (1.48) | 1.45 (1.35) | 0.92 (1.02)
  Day 6 (N=27, 20, 35, 24) | 0.56 (0.75) | 0.85 (1.39) | 1.31 (1.55) | 0.75 (0.90)
  Day 7 (N=27, 21, 34, 22) | 0.48 (0.64) | 0.95 (1.43) | 1.18 (1.57) | 0.59 (0.85)
  Day 8 (N=28, 21, 35, 21) | 0.54 (0.79) | 0.81 (1.29) | 0.94 (1.24) | 0.43 (0.75)

12. Secondary Outcome: Participant's Daily Assessment of Provoked Pain During Post Operative Period: By Treatment Arm
Description: Participants rated pain at 1, 2, 4, 24 and 48 hours after the administration of sugammadex on day of surgery (Day 1), and daily (in the morning) from Day 3 to Day 8. Pain rating was made using an 11-point scale from 0 (no pain) to 10 (severe pain). Separate ratings were made for overall pain at rest, pain when provoked (e.g., due to participant transition from lying to sitting position) and shoulder pain at rest. This measure summarizes the assessment of provoked pain for the study days following the surgery.
Time Frame: Days 2 to 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard NMB and Standard Insufflation Pressure | Standard NMB and Low Insufflation Pressure | Deep NMB and Standard Insufflation Pressure | Deep NMB and Low Insufflation Pressure
Number analyzed (Participants) | 33 | 23 | 40 | 26
score on a scale
  24 hours after sugammadex dose (n=29, 22, 38, 25) | 3.38 (2.37) | 3.27 (2.76) | 3.68 (1.92) | 3.76 (2.47)
  48 hours after sugammadex dose (n=27, 22, 33, 23) | 2.67 (1.96) | 2.14 (2.19) | 2.94 (2.08) | 2.91 (1.83)
  Day 3 (N=22, 20, 30, 17) | 2.23 (1.51) | 2.50 (2.33) | 2.97 (2.11) | 3.24 (2.11)
  Day 4 (N=28, 20, 37, 23) | 2.25 (1.69) | 1.85 (1.95) | 3.05 (2.17) | 1.91 (1.56)
  Day 5 (N=27, 21, 38, 24) | 1.93 (1.54) | 1.90 (1.84) | 2.58 (1.90) | 1.71 (1.46)
  Day 6 (N=27, 20, 35, 24) | 1.70 (1.59) | 1.40 (1.82) | 2.51 (2.06) | 1.42 (1.28)
  Day 7 (N=27, 21, 34, 22) | 1.37 (1.28) | 1.52 (1.66) | 2.21 (2.24) | 1.23 (1.38)
  Day 8 (N=28, 21, 35, 21) | 1.21 (1.34) | 1.38 (1.75) | 1.91 (2.02) | 0.81 (1.08)

13. Secondary Outcome: Participant's Daily Assessment of Shoulder Pain During Post Operative Period: By Treatment Arm
Description: Participants rated pain at 1, 2, 4, 24 and 48 hours after the administration of sugammadex on day of surgery (Day 1), and daily (in the morning) from Day 3 to Day 8. Pain rating was made using an 11-point scale from 0 (no pain) to 10 (severe pain). Separate ratings were made for overall pain at rest, pain when provoked (e.g., due to participant transition from lying to sitting position) and shoulder pain at rest. This measure summarizes the assessment of shoulder pain for the study days following the surgery.
Time Frame: Days 2 to 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard NMB and Standard Insufflation Pressure | Standard NMB and Low Insufflation Pressure | Deep NMB and Standard Insufflation Pressure | Deep NMB and Low Insufflation Pressure
Number analyzed (Participants) | 33 | 23 | 40 | 26
score on a scale
  24 hours after sugammadex dose (n=29, 22, 38, 25) | 1.00 (1.71) | 1.18 (2.15) | 1.05 (1.66) | 1.40 (2.33)
  48 hours after sugammadex dose (n=27, 22, 33, 23) | 0.41 (0.97) | 0.64 (1.22) | 0.76 (1.23) | 0.96 (2.12)
  Day 3 (N=22, 20, 30, 17) | 0.18 (0.50) | 0.80 (1.32) | 0.67 (1.40) | 0.88 (1.76)
  Day 4 (N=28, 20, 37, 23) | 0.32 (1.09) | 0.55 (1.23) | 0.70 (1.60) | 0.61 (1.27)
  Day 5 (N=27, 21, 38, 24) | 0.00 (0.00) | 0.43 (0.81) | 0.68 (1.65) | 0.25 (0.85)
  Day 6 (N=27, 20, 35, 24) | 0.00 (0.00) | 0.15 (0.37) | 0.63 (1.55) | 0.21 (0.83)
  Day 7 (N=27, 21, 34, 22) | 0.00 (0.00) | 0.14 (0.48) | 0.68 (1.63) | 0.23 (0.69)
  Day 8 (N=28, 21, 35, 21) | 0.04 (0.19) | 0.24 (0.44) | 0.66 (1.49) | 0.14 (0.36)

14. Secondary Outcome: Number of Participants Using Pain/Analgesic Medication During Post Operative Period: By Treatment Arm
Description: Post operative use of pain/analgesic medication by participant through Day 8 was recorded.
Time Frame: Up to Day 8
Population: as for outcome 11
Measure: Number; unit: participants using pain medication
Arm/Group | Standard NMB and Standard Insufflation Pressure | Standard NMB and Low Insufflation Pressure | Deep NMB and Standard Insufflation Pressure | Deep NMB and Low Insufflation Pressure
Number analyzed (Participants) | 33 | 23 | 40 | 26
participants using pain medication
  Within 3 hours post surgery | 31 | 21 | 37 | 24
  3 to 24 hours post surgery | 26 | 21 | 38 | 24
  24 to 48 hours post surgery | 26 | 22 | 35 | 23
  Between 48 hours and end of Day 5 | 27 | 20 | 29 | 17
  On Day 6, 7 or 8 | 19 | 14 | 25 | 10

ADVERSE EVENTS:
Time Frame: Up to Day 8
Description: Includes randomized participants with available data who had NMB or pneumoperitoneum for laparoscopic surgery, or received sugammadex. Participants were included in arm corresponding to treatment actually received, which in case of rescue intervention was the post-intervention condition.
Arm/Group | Standard NMB and Standard Insufflation Pressure | Standard NMB and Low Insufflation Pressure | Deep NMB and Standard Insufflation Pressure | Deep NMB and Low Insufflation Pressure
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/23 | 1/40 | 2/26
Other Adverse Events (participants affected / at risk) | 31/33 | 23/23 | 39/40 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard NMB and Standard Insufflation Pressure (N=33) | Standard NMB and Low Insufflation Pressure (N=23) | Deep NMB and Standard Insufflation Pressure (N=40) | Deep NMB and Low Insufflation Pressure (N=26)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard NMB and Standard Insufflation Pressure (N=33) | Standard NMB and Low Insufflation Pressure (N=23) | Deep NMB and Standard Insufflation Pressure (N=40) | Deep NMB and Low Insufflation Pressure (N=26)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (4) | 4 (5) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (11) | 3 (3) | 8 (8) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (6) | 2 (2) | 6 (6) | 3 (3)
Pain (General disorders) | 3 (3) | 3 (4) | 3 (4) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 5 (5) | 3 (3) | 4 (5)
Procedural nausea (Injury, poisoning and procedural complications) | 3 (3) | 1 (2) | 4 (5) | 3 (4)
Procedural pain (Injury, poisoning and procedural complications) | 28 (46) | 19 (34) | 34 (63) | 24 (42)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Wound haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 3 (3) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 8 (8) | 5 (5)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Initial public presentation of the Investigator's results will occur only together with the other sites unless permission is obtained from Sponsor. Sponsor must be able to review all proposed results communications regarding study 45 days prior to submission for publication/presentation. In case of disagreement concerning appropriateness of materials, Investigator and Sponsor must meet to make a good faith effort to discuss/resolve the issues, prior to submission for publication/presentation.